CLINICAL TRIAL: NCT01419951
Title: LAUNCH II: Learning About Activity and Understanding Nutrition for Better Child Health
Brief Title: Launch II: A Pilot Randomized Control Trial of a Clinic and Clinic Plus Home Intervention for Preschool Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008-0666; K24DK059492 (NIH)
Record Dates: First submitted 2011-08-05; First posted 2011-08-18 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Obesity
Keywords: Behavioral treatment; Preschool aged children; Obesity
MeSH Terms: conditions — Obesity | interventions — Ambulatory Care Facilities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Clinic Only Behavioral Intervention (Active Comparator): A 6 month intervention consisting of two phases: Phase I Intensive intervention is 6 sessions delivered in a group-based format in clinic (concurrent parent and child groups) every other week. Phase II Maintenance is 3 monthly clinic visits. Treatment targets 3 components: Dietary education, physical activity and parenting training.
  Interventions: Behavioral: Clinic Only Behavioral Intervention
- Pediatrician Counseling (Active Comparator): A one-time 45 minute visit with a board certified pediatrician that focuses on the AAP guidelines for eating and physical activity for preschool aged children.
  Interventions: Other: Pediatrician Counseling
- Clinic + Home Behavioral Intervention (Experimental): A 6 month intervention consisting of two phases: Phase I Intensive intervention is 12 weekly sessions that alternate between a group-based clinic session (concurrent parent and child groups) and individual home visits. Phase II Maintenance is 12 weeks of every other week visits alternating between clinic and home. Treatment targets 3 components: Dietary education, physical activity and parenting training.
  Interventions: Behavioral: Clinic + Home Behavioral Intervention

INTERVENTIONS:
Behavioral: Clinic + Home Behavioral Intervention — A 6 month intervention consisting of two phases: Phase I Intensive intervention is 12 weekly sessions that alternate between a group-based clinic session (concurrent parent and child groups) and individual home visits. Phase II Maintenance is 12 weeks of every other week visits alternating between clinic and home. Treatment targets 3 components: Dietary education, physical activity and parenting training.
  Arms: Clinic + Home Behavioral Intervention
Other: Pediatrician Counseling — A one-time 45 minute visit with a board certified pediatrician that focuses on the AAP guidelines for eating and physical activity for preschool aged children.
  Arms: Pediatrician Counseling
Behavioral: Clinic Only Behavioral Intervention — A 6 month intervention consisting of two phases: Phase I Intensive intervention is 6 sessions delivered in a group-based format in clinic (concurrent parent and child groups) every other week. Phase II Maintenance is 3 monthly clinic visits. Treatment targets 3 components: Dietary education, physical activity and parenting training.
  Arms: Clinic Only Behavioral Intervention

SUMMARY:
The objective of this project is to pilot test a behavioral intervention that includes a home visit component compared to a clinic only and standard of care for the treatment of obesity in preschool age children. The results of this study will inform the design of a larger randomized control trial.

H1: The clinic + home intervention will result in a significantly greater decrease in BMIz compared to the in clinic only intervention or pediatric standard of care at 6 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* 2 years 0 months to 5 years 11 months of age
* at or above the 95th percentile BMI for age and sex
* have at least one parent with a BMI at or greater than 25
* medical clearance from pediatrician

Exclusion Criteria:

* non-English speaking
* living greater than 50 miles from medical center
* a disability or illness that would preclude engagement in moderate activity
* medical condition/medication associated with weight
* enrolled in another weight management program

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2009-05; Primary Completion 2011-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in BMI z score | Change from Baseline to 6 months
  Body mass index z score

SECONDARY OUTCOMES:
Change in Parent weight loss | Change from baseline to 6 months
Change in Child caloric intake | Change from baseline to 6 months
Change in Home food and activity environment | Change from baseline to 6 months
Change in Child physical activity | Change from baseline to 6 months
Change in Parent-child mealtime interactions | Change from baseline to 6 months
Change in Health related quality of life | Change from baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lori J Stark, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States